CLINICAL TRIAL: NCT03598920
Title: Study of Safety and Efficacy Assessment of Aspiration Therapy for Morbidly Obese Adolescents
Brief Title: Aspiration Therapy for Obese Adolescents
Status: Completed | Type: Observational
Sponsor: University Hospital Ostrava (Other)
Collaborators: University of Ostrava (Other); Vítkovice Hospital Ostrava, Czech Republic (Unknown)
Responsible Party: Sponsor
Other Study IDs: FNO-IK-Aspiration
Record Dates: First submitted 2018-06-13; First posted 2018-07-26 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Obesity, Morbid
Keywords: obesity; bariatric medicine; endoscopy treatment; body composition; Adipokines; Ghrelin; Quality of Life; nutrition status; vitamins
MeSH Terms: conditions — Obesity, Morbid; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AspireAssist: Patients undergoing the endoscopic bariatric procedure using the AsspireAssist device
  Interventions: Device: AsspireAssist
- Nutritional consulting: Patients undergoing nutritional consulting
  Interventions: Other: Nutritional consulting

INTERVENTIONS:
Device: AsspireAssist — Endoscopic bariatric procedure using the AsspireAssist device
  Groups: AspireAssist
Other: Nutritional consulting — Nutritional consulting provided by a specialized consultant.
  Groups: Nutritional consulting

SUMMARY:
Interventional studies devoted to adolescents are relatively rare in the world. This has several reasons. Treatment and research on obesity are centered on advanced forms of obesity in adults, bearing in mind that social and health problems make these patients cope with their condition. Studies on children tend to focus on epidemiology. On the other hand, effective long-term effective treatment is not just for young adults and adolescents. However, appropriate long-term weight reduction methods could help with chronic obesity at the onset of the disease. Here, the ideal scheme at the outset of the disease is to use less invasive endoscopic methods and then use invasive surgical methods at a later age.

The benefit of this study will certainly be to find out the reality of the use of this endoscopic method in young obese individuals, that is, population groups where, according to the WHO and CDC (Centers for Disease Control and Prevention), there has been a rapid increase in the incidence of obesity especially during the last 20 years.

DETAILED DESCRIPTION:
The aim of the project is the testing and research of the impact on metabolism using the approved bariatric method AspireAssist, which is currently used in the adult population. The method has been approved by FDA since 2016. The method involves the introduction of percutaneous endoscopic gastrostomy (PEG) that allows the aspiration of a portion of the food and the control of the size and volume of the food received, even in the unmanaged size and volume of food intake.

Potential participants of the study will undergo an initial examination at the clinical department of pediatric medicine specializing in obesitology at the Vítkovice Hospital Ostrava a.s. In addition to a pediatric and internal examination, a potential patient will be examined by a clinical psychologist for the ability to participate in such a type of study on a long-term basis, and will further assess the degree of patient support and co-operation. Selected participants in the study or their family members will receive informed consent. A study participant is considered to be a participant in the study after consent to his / her inclusion in the study after the informed consent has been signed. The AspireAssist aspiration device is the definitive participation in the study.

Two parts will be monitored within the project. (1) Safety and efficacy will be assessed first in young obese patients for whom the use of bariatric methods is still a question of discussion, especially in surgical methods. (2) The second objective is to monitor the saccharide and lipid metabolism, GI hormones and also the impact of the AspireAssist method on the nutritional status of the adolescents studied.

The patients enrolled in the study are followed for the period of twelve months.

Timetable of the study procedures and controls:

Preoperative examination:

* Demographic data on age, sex, weight, height, smoking
* Assessment of body composition and sampling of blood
* Questionnaires for the quality of Life Examination 3 months postoperatively
* Assessment of body composition and sampling of blood
* Questionnaires for the quality of Life Examination 6 months after surgery
* Assessment of body composition and sampling of blood
* Questionnaires for the quality of Life Examination 12 months after surgery
* Assessment of body composition and sampling of blood
* Questionnaires for the quality of Life

Statistical data processing for statistical evaluation descriptive statistics is used (arithmetical average, standard deflection, frequency tables), X2 test, Fisher's exact test, analysis of variance (ANOVA), calculating of the OR (odds ratio) with 95 % confidence intervals, and logistic regression. Statistical tests are evaluated at the significance level of 5%. Statistical analysis is performed in the "Stata 10" programme. Program EpiData is used for data collection.

ELIGIBILITY:
Inclusion Criteria:

- history of conservative obesity treatments selected according to criteria IFSO (BMI greater than 40 or greater than 35 with comorbidities)

Exclusion Criteria:

* Diabetes Type I.
* blood clotting disorder
* using of Insulin
* psychiatric disorders
* monogenic obesity (Prader-Willi syndrome, mutation of MC4R).
* thyroid disease
* diseases of the digestive system associated with disorders of intestinal absorption
* history of corticosteroid therapy in the past 12 months
* history of bulimia and other eating disorders

Ages: 16 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Adolescents with malignant obesity (BMI> 40) in range BMI 30-50 kg/m2.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Long-term weight reduction assessment in kgs | 12 months
  Evaluation of the success of treatment in terms of long-term weight reduction (difference in body weight in kilograms at the beginning vs. the end of the observation period of 12 months).
Long-term changes of nutritional status | 12 months
  Analysis of the dynamics of changes in nutrition status in adolescents after endoscopic bariatric treatment of obesity (BMI> 30) will be performed. In the study, serum concentrations of the following parameters will be measured: vitamins A, D, E, K, B1, B6, B12, Folic acid and plasma proteins such as albumin, pre albumin, creatinine. The measurements will be performed before the planned intervention and then in intervals at 3, 6 and 12 months after the procedure. The results will be presented in mmol/L.

SECONDARY OUTCOMES:
Changes in serum levels of adipose tissue hormones | 12 months
  Analysis of the dynamics of changes in serum levels of adipose tissue hormones (Leptin, Adiponectin) in adolescents after endoscopic bariatric treatment of obesity (BMI> 30) will be performed. Points of measurements: before the planned intervention and then in intervals of 3, 6 and 12 months after procedure.
Changes in serum levels of lipids | 12 months
  Analysis of the dynamics of changes in serum levels of lipids in adolescents after endoscopic bariatric treatment of obesity (BMI> 30) will be performed. In the study, serum concentrations of the following lipids will be measured: triacylglycerols, total cholesterol, high-density lipoprotein, low-density lipoprotein cholesterol, Apo D and Apo E, FGF 21, FGF19, FXR receptor, Omentin 1. The measurements will be performed before the planned intervention and then in intervals at 3, 6 and 12 months after the procedure. The results will be presented in mmol/L.
Changes in serum levels GI hormones and saccharide metabolism | 12 months
  Analysis of the dynamics of changes in serum levels of usual panel of GI hormones in adolescents after endoscopic bariatric treatment of malignant obesity (BMI> 35) will be performed. The following serum levels markers of bone resorption and formation will be assessed: fasting glycaemia, insulin and hemoglobin A1C, C-peptide, acylated ghrelin, GLP-1, GIP, PYY. The measurements will be performed before the planned intervention and then in intervals at 3, 6 and 12 months after the procedure. The results will be presented in mmol/L.
IWQOL Questionnaire evaluation | 12 months
  Evaluation of effects of endoscopic bariatric interventions on quality of life will be performed by using the IWQOL questionnaire. Improvement from baseline quality of life as measured by standardized IWQOL patient questionnaire (http://www.qualityoflifeconsulting.com/iwqol-lite.html) intended to measure the patient health status.
SF-36 Questionnaire evaluation | 12 months
  Evaluation of effects of different types of bariatric interventions on the quality of life will be performed using the SF-36 questionnaire. Improvement from baseline quality of life as measured by standardized SF-36 patient questionnaire intended to measure the patient health status.

CONTACTS AND LOCATIONS:
Overall Officials: Evžen Machytka, MD,Ph.D., Principal Investigator — University Hospital Ostrava
Locations (3):
- Czechia (3):
  - Ostrava University, Ostrava, Moravian-Silesian Region
  - Vítkovice Hospital Ostrava, Ostrava, Moravian-Silesian Region
  - University Hospital Ostrava, Ostrava, Moravian-Silesian Region

IPD SHARING:
Plan to Share IPD: Undecided
The investigators have not decided to share IPD with other researchers.

REFERENCES:
- [Background] Nystrom M, Machytka E, Noren E, Testoni PA, Janssen I, Turro Homedes J, Espinos Perez JC, Turro Arau R. Aspiration Therapy As a Tool to Treat Obesity: 1- to 4-Year Results in a 201-Patient Multi-Center Post-Market European Registry Study. Obes Surg. 2018 Jul;28(7):1860-1868. doi: 10.1007/s11695-017-3096-5. PMID 29388050
- [Background] Sullivan S, Edmundowicz SA, Thompson CC. Endoscopic Bariatric and Metabolic Therapies: New and Emerging Technologies. Gastroenterology. 2017 May;152(7):1791-1801. doi: 10.1053/j.gastro.2017.01.044. Epub 2017 Feb 10. PMID 28192103
- [Background] Abu Dayyeh BK, Edmundowicz S, Thompson CC. Clinical Practice Update: Expert Review on Endoscopic Bariatric Therapies. Gastroenterology. 2017 Mar;152(4):716-729. doi: 10.1053/j.gastro.2017.01.035. Epub 2017 Jan 29. PMID 28147221
- [Background] Kumar N, Sullivan S, Thompson CC. The role of endoscopic therapy in obesity management: intragastric balloons and aspiration therapy. Diabetes Metab Syndr Obes. 2017 Jul 6;10:311-316. doi: 10.2147/DMSO.S95118. eCollection 2017. PMID 28740414
- [Background] Sullivan S. Aspiration Therapy for Obesity. Gastrointest Endosc Clin N Am. 2017 Apr;27(2):277-288. doi: 10.1016/j.giec.2016.12.001. PMID 28292406
- [Background] Kumbhari V, Okolo PI III. Editorial: Aspiration Therapy for Weight Loss: Is the Squeeze worth the Juice? Am J Gastroenterol. 2017 Mar;112(3):458-589. doi: 10.1038/ajg.2017.2. PMID 28270668
- [Background] ASGE Bariatric Endoscopy Task Force; ASGE Technology Committee; Abu Dayyeh BK, Edmundowicz SA, Jonnalagadda S, Kumar N, Larsen M, Sullivan S, Thompson CC, Banerjee S. Endoscopic bariatric therapies. Gastrointest Endosc. 2015 May;81(5):1073-86. doi: 10.1016/j.gie.2015.02.023. Epub 2015 Mar 28. No abstract available. PMID 25828245
- [Background] Devault KR. Could aspiration therapy for obesity be an effective and safe alternative to traditional bariatric surgery? Gastroenterology. 2013 Dec;145(6):1188-90. doi: 10.1053/j.gastro.2013.10.038. No abstract available. PMID 24409479
- [Background] Sullivan S, Stein R, Jonnalagadda S, Mullady D, Edmundowicz S. Aspiration therapy leads to weight loss in obese subjects: a pilot study. Gastroenterology. 2013 Dec;145(6):1245-52.e1-5. doi: 10.1053/j.gastro.2013.08.056. Epub 2013 Sep 6. PMID 24012983
- [Background] Forssell H, Noren E. A novel endoscopic weight loss therapy using gastric aspiration: results after 6 months. Endoscopy. 2015 Jan;47(1):68-71. doi: 10.1055/s-0034-1378097. Epub 2014 Sep 30. PMID 25268305